CLINICAL TRIAL: NCT05939726
Title: A Phase II, Randomised Controlled Trial to Evaluate the Efficacy and Safety of Moisturising Creams With or Without Palm-oil-derived Vitamin E Concentrate in Addition to Urea-based Cream or Urea-based Cream Alone in Capecitabine-associated Palmar-Plantar Erythrodysesthesia (ECaPPE)
Brief Title: Efficacy and Safety of Moisturising Cream With or Without Vitamin E and Urea Cream in Palmar-plantar Erythrodysesthesia
Acronym: ECaPPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarawak General Hospital (Other)
Collaborators: Avantsar Sdn. Bhd. (Unknown); Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Voon Pei Jye, Medical Oncologist, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRC005-ECaPPE
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Palmar-Plantar Erythrodysesthesia; Palmar-Plantar Erythrodysesthesia Due to Cytotoxic Therapy
Keywords: Palmar-Plantar Erythrodysesthesia; Cytotoxic therapy; Capecitabine; Vitamin E; Tocotrienol; Tocopherol; Topical applications; Randomised controlled trial; Urea cream; Hand-foot syndrome; Supportive care
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The use of the investigational creams, i.e. moisturising creams with or without vitamin E concentrate will be double-blinded. Both creams will be the same in colour, texture, packaging, and labelling. The patients, investigators, and blinded study personnel will blinded the patients' assignment of the investigational creams. On the other hand, the use of urea cream will be open-labelled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moisturising Cream with Vitamin E and Urea Cream (Experimental): Participants who are randomised in this arm will receive a moisturising cream containing palm-oil-derived vitamin E concentrate for external application on both palms and soles, in addition to urea-based cream as the standard of care for PPE management. They will be required to apply the investigational cream first, followed by the urea-based cream, at least two times a day.
  Interventions: Other: Moisturising cream with vitamin E concentrate; Other: Urea cream
- Moisturising Cream without Vitamin E and Urea Cream (Experimental): Participants who are randomised to this arm will receive a basic or plain moisturising cream without Vitamin E for external application on both palms and soles, in addition to urea-based cream as the standard of care for PPE management. They will be required to apply the investigational cream first, followed by the urea-based cream, at least two times a day.
  Interventions: Other: Moisturising cream without vitamin E concentrate; Other: Urea cream
- Urea Cream Only (Active Comparator): Participants who are randomised to this arm will receive urea-based cream only as the standard of care for PPE management. They will be required to use the urea cream at least twice a day.
  Interventions: Other: Urea cream

INTERVENTIONS:
Other: Moisturising cream with vitamin E concentrate — The vitamin E moisturising cream contains 3% w/w of palm-oil-derived vitamin E concentrate, consisting of the following isomers: alpha-tocopherol, alpha-tocotrienol, beta-tocotrienol, gamma-tocotrienol, and delta-tocotrienol. This formula provides a total of 1.2g tocotrienols per 100g product.
  Arms: Moisturising Cream with Vitamin E and Urea Cream
Other: Moisturising cream without vitamin E concentrate — This moisturising cream is a similar moisturising cream but without the addition of the vitamin E concentrate
  Arms: Moisturising Cream without Vitamin E and Urea Cream
Other: Urea cream — Urea cream (10%w/w) is used as the standard of care for PPE.

SUMMARY:
This is a single-centre, phase II, three-arm, randomised controlled trial to evaluate the efficacy and safety of a cosmetic moisturising cream containing palm-oil-derived vitamin E concentrate or a similar moisturising cream without the vitamin E concentrate in addition to urea-based cream, or urea-based cream alone (1:1:1) in patients who are receiving capecitabine-based cancer therapy and develop capecitabine-associated PPE of NCI-CTCAE grade 1.

DETAILED DESCRIPTION:
In this study, cancer patients from Sarawak General Hospital who are receiving capecitabine-based therapy and develop PPE of NCI-CTCAE grade 1 will be recruited and randomised 1:1:1 to three study arms. The participants who are randomised to treatment arms will receive moisturising creams with or without palm-oil-derived vitamin E concentrate, in addition to urea-based cream for external application on palms and soles. Participants who are randomised to the control arm will be required to use urea-based cream only.

Both patients and investigators will be blinded to the investigational cream assignment i.e., double-blind. However, blinding will not be applicable to the use of urea cream i.e., open-label. The patients will need to use the cream(s) at least two times a day for nine to eighteen weeks or equivalent to three to six treatment cycles of capecitabine. At week-9, the patients who are planned to continue capecitabine therapy and do not develop PPE of grade 2/3 will continue to receive the study treatments for additional nine weeks or equivalent to three treatment cycles of capecitabine (extended period).

The patients will be assessed for their PPE grading, symptoms, dermatological quality of life, pain score, and adverse events at the end of each capecitabine treatment cycle at the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above
2. Able to give written consent freely
3. Receiving capecitabine at least 1 dose, as monotherapy or in combination therapy
4. Receiving urea-based cream
5. Developed PPE of NCI-CTCAE grade 1
6. Have at least three cycles of chemotherapy to complete
7. Life expectancy ≥ 6 months
8. ECOG≤2

Exclusion Criteria:

1. Unable to understand the information sheet and informed consent form
2. Allergy history towards vitamin E and its isoforms or any components of the investigational products
3. Unable to tolerate urea-based products
4. Other pre-existing dermatological diseases or conditions that may interfere the evaluation of PPE
5. PPE complicated with infection
6. Receiving other agent(s) that are known to cause PPE or hand- foot syndrome and hand-foot skin reactions
7. Receiving long-term topical or systemic steroid treatment (except as part of pre-or post-medications of chemotherapy regime)
8. Pregnant or lactating mother
9. Participating in another interventional trial
10. Refuses to interrupt his/her usual care
11. Anticipated inability to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Palmar-plantar erythrodysesthesia (PPE) resolution | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Number of participants who have resolved PPE (NCI-CTCAE grade 1 to 0)

SECONDARY OUTCOMES:
Palmar-plantar erythrodysesthesia (PPE) worsening | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Number of participants who have worsened PPE (NCI-CTCAE grade 1 to 2/3)
Time-to-PPE resolution | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Time-to-PPE resolution via patient self-reported symptoms in standardised diary
Time-to-PPE worsening | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Time-to-PPE worsening via patient self-reported symptoms in standardised diary
Dermatology Life Quality Index (0 - 30) | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  The Dermatology Life Quality Index (DLQI) consists of 10 questions, and each question is assigned a score (0 to 3). The total score ranges from 0 to 30, with higher scores indicating greater impairment in the individual's quality of life.
Pain score (numerical scale of 1 to 10) | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  The pain score is assessed using a 1-10 numeric rating pain scale, where 1 represents no pain at all, and 10 is the worst pain.
Overall adverse events | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Frequency of overall adverse events
Dermatology-related adverse events | At Day 22, Day 43, Day 64, and Day 127 of cream treatment
  Frequency of dermatology-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Pei Jye Voon, M.D, Principal Investigator — Sarawak General Hospital
Locations (1):
- Sarawak General Hospital, Kuching, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gressett SM, Stanford BL, Hardwicke F. Management of hand-foot syndrome induced by capecitabine. J Oncol Pharm Pract. 2006 Sep;12(3):131-41. doi: 10.1177/1078155206069242. PMID 17022868
- [Background] Nikolaou V, Syrigos K, Saif MW. Incidence and implications of chemotherapy related hand-foot syndrome. Expert Opin Drug Saf. 2016 Dec;15(12):1625-1633. doi: 10.1080/14740338.2016.1238067. Epub 2016 Oct 8. PMID 27718746
- [Background] Kwakman JJM, Elshot YS, Punt CJA, Koopman M. Management of cytotoxic chemotherapy-induced hand-foot syndrome. Oncol Rev. 2020 May 13;14(1):442. doi: 10.4081/oncol.2020.442. eCollection 2020 Feb 18. PMID 32431787
- [Background] Lou Y, Wang Q, Zheng J, Hu H, Liu L, Hong D, Zeng S. Possible Pathways of Capecitabine-Induced Hand-Foot Syndrome. Chem Res Toxicol. 2016 Oct 17;29(10):1591-1601. doi: 10.1021/acs.chemrestox.6b00215. Epub 2016 Sep 28. PMID 27631426
- [Background] Milano G, Etienne-Grimaldi MC, Mari M, Lassalle S, Formento JL, Francoual M, Lacour JP, Hofman P. Candidate mechanisms for capecitabine-related hand-foot syndrome. Br J Clin Pharmacol. 2008 Jul;66(1):88-95. doi: 10.1111/j.1365-2125.2008.03159.x. Epub 2008 Mar 13. PMID 18341672
- [Background] Zhang RX, Wu XJ, Lu SX, Pan ZZ, Wan DS, Chen G. The effect of COX-2 inhibitor on capecitabine-induced hand-foot syndrome in patients with stage II/III colorectal cancer: a phase II randomized prospective study. J Cancer Res Clin Oncol. 2011 Jun;137(6):953-7. doi: 10.1007/s00432-010-0958-9. Epub 2010 Nov 27. PMID 21113620
- [Background] Hofheinz RD, Gencer D, Schulz H, Stahl M, Hegewisch-Becker S, Loeffler LM, Kronawitter U, Bolz G, Potenberg J, Tauchert F, Al-Batran SE, Schneeweiss A. Mapisal Versus Urea Cream as Prophylaxis for Capecitabine-Associated Hand-Foot Syndrome: A Randomized Phase III Trial of the AIO Quality of Life Working Group. J Clin Oncol. 2015 Aug 1;33(22):2444-9. doi: 10.1200/JCO.2014.60.4587. Epub 2015 Jun 29. PMID 26124485
- [Background] Wolf SL, Qin R, Menon SP, Rowland KM Jr, Thomas S, Delaune R, Christian D, Pajon ER Jr, Satele DV, Berenberg JL, Loprinzi CL; North Central Cancer Treatment Group Study N05C5. Placebo-controlled trial to determine the effectiveness of a urea/lactic acid-based topical keratolytic agent for prevention of capecitabine-induced hand-foot syndrome: North Central Cancer Treatment Group Study N05C5. J Clin Oncol. 2010 Dec 10;28(35):5182-7. doi: 10.1200/JCO.2010.31.1431. Epub 2010 Nov 8. PMID 21060036
- [Background] Hoesly FJ, Baker SG, Gunawardane ND, Cotliar JA. Capecitabine-induced hand-foot syndrome complicated by pseudomonal superinfection resulting in bacterial sepsis and death: case report and review of the literature. Arch Dermatol. 2011 Dec;147(12):1418-23. doi: 10.1001/archdermatol.2011.320. PMID 22184763
- [Background] Kara IO, Sahin B, Erkisi M. Palmar-plantar erythrodysesthesia due to docetaxel-capecitabine therapy is treated with vitamin E without dose reduction. Breast. 2006 Jun;15(3):414-24. doi: 10.1016/j.breast.2005.07.007. Epub 2005 Sep 26. PMID 16188440
- [Background] Yamamoto D, Yamamoto C, Iwase S, Kuroda Y, Odagiri H, Nagumo Y. Efficacy of Vitamin E Treatment for Hand-Foot Syndrome in Patients Receiving Capecitabine. Breast Care (Basel). 2010;5(6):415-416. doi: 10.1159/000322660. Epub 2010 Nov 26. No abstract available. PMID 21494409
- [Background] Bozkurt Duman B, Kara B, Oguz Kara I, Demiryurek H, Aksungur E. Hand-foot syndrome due to sorafenib in hepatocellular carcinoma treated with vitamin E without dose modification; a preliminary clinical study. J BUON. 2011 Oct-Dec;16(4):759-64. PMID 22331734